CLINICAL TRIAL: NCT06916832
Title: Evaluation of the Impact of Implementing a Patient Blood Management Protocol on the Transfusion Rate in Delivery Hemorrhage
Brief Title: Evaluation of a Patient Blood Management Protocol Impact on the Transfusion Rate in Delivery Hemorrhage
Acronym: PALOMA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-CHITS-018
Record Dates: First submitted 2025-03-11; First posted 2025-04-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Delivery Hemorrhage
Keywords: Delivery hemorrhage; Pregnancy; Blood transfusion; Patient blood management; Iron supplementation; Gestational anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before protocol implementation: pregnant women who did not use the patient blood management protocol during their pregnancy. In other words, women who gave birth in 2023 and 2024.
- After protocol implementation: pregnant women who benefited from the patient blood management protocol during their pregnancy. In other words, women who gave birth in 2025.

SUMMARY:
According to the WHO, anemia is one of the ten most serious health problems in the world. During pregnancy, it affects 42% of women worldwide and 25% in France. It is associated with an increased risk of perinatal morbidity and mortality, and recourse to blood transfusion. The blood transfusion is itself also a source of thromboembolic morbidity and mortality, infectious diseases and pulmonary pathologies. In addition, the risk of hemorrhage, particularly during delivery, is inherent to all pregnancies and difficult to predict.

Since 2010, the WHO has defined the rational use of blood products as the 4th global priority, and the need for countries to reduce blood transfusion. It introduces the concept of Patient Blood Management (PBM). This is a set of measures designed to manage anemia and bleeding in surgical patients, while avoiding the need for transfusion. These measures include preoperative screening for anemia and martial deficiency, iron and vitamin supplementation, intraoperative bleeding control and optimization of postoperative blood balance. Recommended by several national programs, PBM has developed rapidly in orthopedic and cardiac surgery, where numerous studies have demonstrated its effectiveness, particularly in terms of transfusion savings. In obstetrics, however, the implementation of PBM remains less widespread, notably due to the difficulty of getting teams on board, and the absence of protocolization.

However, given the high prevalence of anemia in pregnant women, and the inherent risk of hemorrhage in all deliveries with potential recourse to blood transfusion, personalized optimization of PBM is a major challenge in obstetrics.

The PBM is currently being implemented in routine practice in the CHITS maternity department, in line with recommendations.

In this context, our research aims to assess the impact of this new approach. Our main hypothesis is that implementation of a PBM protocol would reduce the rate of transfusion in delivery hemorrhage.

DETAILED DESCRIPTION:
From 1 January 2023 to 31 December 2025, the investigators conducted a single-center, before-and-after study at the maternity unit of the Sainte Musse hospital in Toulon (level IIB maternity unit). This is a retrospective observational study with a retrospective section covering the period before the implementation of the PBM protocol between 1 January 2023 and 31 December 2024. Then a prospective part covering the period after the implementation of the PBM protocol, from 1 January 2025 to 31 December 2025.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has had a delivery hemorrhage, whatever the mode of delivery

Exclusion Criteria:

* Minor
* Under legal protection
* Hemoglobinopathies
* Patient's refusal to participate in research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who suffered a delivery hemorrhage during childbirth,in the maternity ward of Hôpital Sainte Musse
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
RGC transfusion rate | 24 hours postpartum
  Comparison of the RGC transfusion rate over the length of stay following delivery hemorrhage between the 2 periods (before and after PBM implementation).

SECONDARY OUTCOMES:
Number of RGCs transfused during the first 24 hours postpartum | 24 hours postpartum
Prescription of intra-venous iron during pregnancy | 24 hours postpartum
  Number of patients with at least one prescription for IV iron during pregnancy.
Hemoglobin level at hospital discharge | Day 7 postpartum
  average hemoglobin level at discharge (before vs. after protocol implementation)
Treatments for the management of delivery haemorrhage. | Day 7 postpartum
  Number of patients who will use the following treatments: Tranexamic acid, Fibrinogen, Syntocinon, Nalador, FFP transfusion, DA-RU (artificial delivery, uterine revision), surgical treatment, bakri balloon

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine SLEHOHER-LHERIAU, MD, Study Director — Centre Intercommunal Toulon-La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal de Toulon-La Seyne sur mer, Toulon, VAR, France

IPD SHARING:
Plan to Share IPD: No